CLINICAL TRIAL: NCT06960720
Title: Lifting More Than Weights: Feasibility of Implementing a Resistance Exercise Program Across Socioeconomic Groups for Cancer-Related Fatigue Management
Brief Title: Lifting More Than Weights: Resistance Exercise Program Across Socioeconomic Groups for Cancer-Related Fatigue Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Megan Clark, Associate Professor, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2501103633
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Fatigue
Keywords: Strength After Breast Cancer; Allostatic load; Cancer Related Fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength After Breast Cancer (SABC) Lower SES (Active Comparator): Strength after Breast Cancer (SABC) is an evidence-based exercise program that improves body composition, body image, strength, and upper body using initial supervised sessions followed by unsupervised sessions with follow-up as needed.
  Interventions: Other: Resistance Exercises
- Strength After Breast Cancer (SABC) Higher SES (Active Comparator): Strength after Breast Cancer (SABC) is an evidence-based exercise program that improves body composition, body image, strength, and upper body using initial supervised sessions followed by unsupervised sessions with follow-up as needed.
  Interventions: Other: Resistance Exercises

INTERVENTIONS:
Other: Resistance Exercises — Twice-weekly resistance exercises completed in 45 minutes using resistance bands and a physical therapy workout plan.

SUMMARY:
The long-term goal of this project is to improve the implementation of tailored resistance exercise interventions for Appalachian breast cancer survivors. To achieve this goal, the primary objective is to enhance the understanding of how biological, psychological, and social factors interact to influence readiness for behavior change around resistance exercise in this unique population. The primary aim is to evaluate the feasibility of delivering the Strength After Breast Cancer (SABC) program, focusing on how socioeconomic status (SES) and allostatic load (AL) scores influence adherence and dropout rates. The Investigators will also further examine how self-efficacy, outcome expectations, and social support influence behavior change related to resistance exercise participation. The central hypothesis is that participants with lower SES will report geographic or financial constraints, receive reduced support from family or peers, have low confidence in their ability to exercise, and demonstrate lower adherence rates.

Participants will:

* Use a clear, step-by-step guide for safe, progressive strength training using a resistance exercise program tailored specifically for breast cancer survivors for a duration of 3 months
* Keep an exercise log and complete questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed Breast Cancer; any tumor molecular subtype can be enrolled.
* Subjects must have been diagnosed with non-metastatic breast cancer, defined as stage 0, I, II, or III (according to the American Joint Committee on Cancer Tumor, Node, Metastasis staging system), and must be between one and three years post-diagnosis at the time of enrollment. With treatment being received from the West Virginia University (WVU) Cancer Institute.
* Any severity or report of fatigue. This can be done through a subjective report documented by any healthcare professional or through a screening tool like the enhanced distress thermometer.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Subjects who are pregnant (first or second trimester) or breastfeeding must receive additional approval from their obstetrics and gynecology physician for participation. Only individuals with a singleton pregnancy (no multiple gestations) will be eligible for participation. Pregnant participants must be in their first or second trimester at the time of enrollment to ensure they can complete the full three-month program before childbirth. Multiple gestations are associated with higher risks of pregnancy complications, increased physical limitations, and a greater likelihood of preterm delivery, which may prevent completion of the program.

Exclusion Criteria:

* Male biological gender. Males will be excluded from the study due to the rarity of male breast cancer and the variability gender creates on AL scores.
* Subjects with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, active alcoholism, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with pregnancy beyond the second trimester at the time of enrollment, as later stages of pregnancy may prevent completion of the full three-month program.
* Subjects who are pregnant with multiple gestations (e.g., twins, triplets, or higher-order pregnancies) due to the increased risk of pregnancy-related complications, physical limitations, and the likelihood of preterm delivery, which may interfere with program completion.
* Subjects whose self-reported household income is above or below the median household income in Appalachia ($61,688) and for whom the target enrollment of 30 participants in that respective SES group (higher or lower) has already been met at the time of screening, as representation of both SES groups is required for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Dropout Rate - Lower SES | 3 Months
  Percentage of participants in the lower SES group who drop out of the program
Dropout Rate - Higher SES | 3 Months
  Percentage of participants in the higher SES group who drop out of the program
Overall Dropout Rate | 3 Months
  Percentage of participants who drop out of the program.

SECONDARY OUTCOMES:
Adherence Rate - Lower SES | 3 Months
  Percentage of participants in the lower SES group completing ≥ 75% of intervention activities and all scheduled assessments.
Adherence Rate - Higher SES | 3 Months
  Percentage of participants in the higher SES group completing ≥ 75% of intervention activities and all scheduled assessments
Overall Adherence Rate | 3 Months
  Percentage of participants completing ≥ 75% of intervention activities and all scheduled assessments.

OTHER OUTCOMES:
FACIT-F - (Lower SES) | Baseline to 3 Month follow up
  Change in score of fatigue will be measured using the Functional Assessment of Chronic Illness-Fatigue (FACIT-F), fatigue subscale. This is a 13-item subscale of the FACIT-F questionnaire in which a higher score indicates less fatigue. Scores range from 0-52.
FACIT-F - (Higher SES) | Baseline to 3 Month follow up
  Change in score of fatigue will be measured using the Functional Assessment of Chronic Illness-Fatigue (FACIT-F), fatigue subscale. This is a 13-item subscale of the FACIT-F questionnaire in which a higher score indicates less fatigue. Scores range from 0-52.
FACIT-F - Overall Change in Score | Baseline to 3 Month follow up
  Change in score of fatigue will be measured using the Functional Assessment of Chronic Illness-Fatigue (FACIT-F), fatigue subscale. This is a 13-item subscale of the FACIT-F questionnaire in which a higher score indicates less fatigue. Scores range from 0-52.
Allostatic Load (AL) Score- (Lower SES) | Baseline to 3 Month Follow Up
  Change in Allostatic Load score. AL score calculations will occur using cardiovascular, metabolic, and immune system biomarkers in the electronic health record (EHR). AL will be calculated by summing the number of biomarkers in the highest-risk quartile according using a range from 0 (low AL) to 10 (high AL).
Allostatic Load (AL) Score - (Higher SES) | Baseline to 3 Month Follow Up
  Change in Allostatic Load score. AL score calculations will occur using cardiovascular, metabolic, and immune system biomarkers in the electronic health record (EHR). AL will be calculated by summing the number of biomarkers in the highest-risk quartile according using a range from 0 (low AL) to 10 (high AL).
Allostatic Load (AL) Score - Overall Change in score | Baseline to 3 Month Follow Up
  Change in Allostatic Load score. AL score calculations will occur using cardiovascular, metabolic, and immune system biomarkers in the electronic health record (EHR). AL will be calculated by summing the number of biomarkers in the highest-risk quartile according using a range from 0 (low AL) to 10 (high AL).
Stages of Change Exercise Continuous Measure - (Lower SES) | Baseline to 3 Month Follow Up
  Change in the Stages of Change Exercise Continuous Measure Score. This is a self-administered 24 item questionnaire to assess an individual's readiness to engage in regular physical activity. The items are categorized into different stages of readiness: Precontemplation, Contemplation, Preparation, Action, and Maintenance. Each item is rated on a Likert-type scale, ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). There are stage scores (sum the responses for items within each stage) and a total score (sum the stage scores to get an overall readiness score). Higher scores in stages indicate a higher level of readiness of the participants.
Stages of Change Exercise Continuous Measure- (Higher SES) | Baseline to 3 Month Follow Up
  Change in the Stages of Change Exercise Continuous Measure Score. This is a self-administered 24 item questionnaire to assess an individual's readiness to engage in regular physical activity. The items are categorized into different stages of readiness: Precontemplation, Contemplation, Preparation, Action, and Maintenance. Each item is rated on a Likert-type scale, ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). There are stage scores (sum the responses for items within each stage) and a total score (sum the stage scores to get an overall readiness score). Higher scores in stages indicate a higher level of readiness of the participants.
Stages of Change Exercise Continuous Measure- Overall Change in Score | Baseline to 3 Month Follow Up
  Change in the Stages of Change Exercise Continuous Measure Score. This is a self-administered 24 item questionnaire to assess an individual's readiness to engage in regular physical activity. The items are categorized into different stages of readiness: Precontemplation, Contemplation, Preparation, Action, and Maintenance. Each item is rated on a Likert-type scale, ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). There are stage scores (sum the responses for items within each stage) and a total score (sum the stage scores to get an overall readiness score). Higher scores in stages indicate a higher level of readiness of the participants.
Self-Efficacy for Exercise - (Lower SES) | Baseline to 3 Month Follow Up
  Change in score for the Self-Efficacy for Exercise (SEE) Scale. This scale is used to assess an individual's confidence in their ability to engage in regular physical activity. It is a 9-item self-administered questionnaire. Each item is rated on a 11-point Likert scale (0 = Not confident at all to 10 = Very confident). Higher scores indicate greater self-efficacy for exercise.
Self-Efficacy for Exercise - (Higher SES) | Baseline to 3 Month Follow Up
  Change in score for the Self-Efficacy for Exercise (SEE) Scale. This scale is used to assess an individual's confidence in their ability to engage in regular physical activity. It is a 9-item self-administered questionnaire. Each item is rated on a 11-point Likert scale (0 = Not confident at all to 10 = Very confident). Higher scores indicate greater self-efficacy for exercise.
Self-Efficacy for Exercise - Overall Change in Score | Baseline to 3 Month Follow Up
  Change in score for the Self-Efficacy for Exercise (SEE) Scale. This scale is used to assess an individual's confidence in their ability to engage in regular physical activity. It is a 9-item self-administered questionnaire. Each item is rated on a 11-point Likert scale (0 = Not confident at all to 10 = Very confident). Higher scores indicate greater self-efficacy for exercise.
Bellarmine Norton Assessment Tool (BNAT) Score - (Lower SES) | Baseline to 3 Month Follow Up
  Change in BNAT score. This is a clinical tool designed to measure physical function in individuals with cancer. It includes both self-reported and objective physical performance components. Each component of the BNAT is scored individually, and these scores are then combined to produce the total BNAT score. Scoring process: - Self-Reported Physical Activity: Rated on a Likert scale (e.g., 1 to 5), where higher scores indicate higher levels of physical activity. - Objective Tests: 2-Minute Step Test: The number of steps is converted into a score (e.g., 1 to 5); 30-Second Sit to Stand: The number of cycles is converted into a score (e.g., 1 to 5); Timed Arm Curl: The number of curls is converted into a score (e.g., 1 to 5); Timed Up and Go (TUG): The time taken is converted into a score (e.g., 1 to 5), with lower times indicating better performance.
  - Total BNAT Score: The total score ranges from 1 to 25, with higher scores indicating higher physical functioning.
Bellarmine Norton Assessment Tool (BNAT) Score - (Higher SES) | Baseline to 3 Month Follow Up
  Change in BNAT score. This is a clinical tool designed to measure physical function in individuals with cancer. It includes both self-reported and objective physical performance components. Each component of the BNAT is scored individually, and these scores are then combined to produce the total BNAT score. Scoring process: - Self-Reported Physical Activity: Rated on a Likert scale (e.g., 1 to 5), where higher scores indicate higher levels of physical activity. - Objective Tests: 2-Minute Step Test: The number of steps is converted into a score (e.g., 1 to 5); 30-Second Sit to Stand: The number of cycles is converted into a score (e.g., 1 to 5); Timed Arm Curl: The number of curls is converted into a score (e.g., 1 to 5); Timed Up and Go (TUG): The time taken is converted into a score (e.g., 1 to 5), with lower times indicating better performance.
  - Total BNAT Score: The total score ranges from 1 to 25, with higher scores indicating higher physical functioning.
Bellarmine Norton Assessment Tool (BNAT) Score - Overall Change in Score | Baseline to 3 Month Follow Up
  Change in BNAT score. This is a clinical tool designed to measure physical function in individuals with cancer. It includes both self-reported and objective physical performance components. Each component of the BNAT is scored individually, and these scores are then combined to produce the total BNAT score. Scoring process: - Self-Reported Physical Activity: Rated on a Likert scale (e.g., 1 to 5), where higher scores indicate higher levels of physical activity. - Objective Tests: 2-Minute Step Test: The number of steps is converted into a score (e.g., 1 to 5); 30-Second Sit to Stand: The number of cycles is converted into a score (e.g., 1 to 5); Timed Arm Curl: The number of curls is converted into a score (e.g., 1 to 5); Timed Up and Go (TUG): The time taken is converted into a score (e.g., 1 to 5), with lower times indicating better performance.
  - Total BNAT Score: The total score ranges from 1 to 25, with higher scores indicating higher physical functioning.
Grip Strength - (Lower SES) | Baseline to 3 Month Follow Up
  Change in Grip strength will be measured using the Jamar hand-held dynamometer which measures in pounds (up to 200 pounds). Higher recorded pounds equal a greater grip strength.
Grip Strength - (Higher SES) | Baseline to 3 Month Follow Up
  Change in grip strength will be measured using the Jamar hand-held dynamometer which measures in pounds (up to 200 pounds). Higher recorded pounds equal a greater grip strength.
Grip Strength - Overall Change in Score | Baseline to 3 Month Follow Up
  Change in grip strength will be measured using the Jamar hand-held dynamometer which measures in pounds (up to 200 pounds). Higher recorded pounds equal a greater grip strength.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core (EORTC QLQ-C30) - (Lower SES) | Baseline to 3 Month Follow Up
  Change in score for the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core (EORTC QLQ-C30). This is a specialized questionnaire designed for cancer patients. It consists of 30 items that evaluate various dimensions of health and well-being, including: Physical Functioning, Role Functioning, Emotional Functioning, Cognitive Functioning, Social Functioning, Global Health Status/Quality of Life, Symptom Scales. In scoring, 28 items are rated on a 4-point scale (1 = Not at all to 4 = Very much), and the last two items use a 7-point scale (1 = Very Poor to 7 = Excellent). Raw scores are linearly transformed to a 0-100 scale. For functional scales and the global health status/QoL scale, higher scores represent better functioning or quality of life. For symptom scales/items, higher scores indicate more severe symptoms.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core (EORTC QLQ-C30) - (Higher SES) | Baseline to 3 Month Follow Up
  Change in score for the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core (30EORTC QLQ-C30). This is a specialized questionnaire designed for cancer patients. It consists of 30 items that evaluate various dimensions of health and well-being, including: Physical Functioning, Role Functioning, Emotional Functioning, Cognitive Functioning, Social Functioning, Global Health Status/Quality of Life, Symptom Scales. In scoring, 28 items are rated on a 4-point scale (1 = Not at all to 4 = Very much), and the last two items use a 7-point scale (1 = Very Poor to 7 = Excellent). Raw scores are linearly transformed to a 0-100 scale. For functional scales and the global health status/QoL scale, higher scores represent better functioning or quality of life. For symptom scales/items, higher scores indicate more severe symptoms.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core (EORTC QLQ-C30) - Overall Change in Score | Baseline to 3 Month Follow Up
  Change in score for the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core (30EORTC QLQ-C30). This is a specialized questionnaire designed for cancer patients. It consists of 30 items that evaluate various dimensions of health and well-being, including: Physical Functioning, Role Functioning, Emotional Functioning, Cognitive Functioning, Social Functioning, Global Health Status/Quality of Life, Symptom Scales. In scoring, 28 items are rated on a 4-point scale (1 = Not at all to 4 = Very much), and the last two items use a 7-point scale (1 = Very Poor to 7 = Excellent). Raw scores are linearly transformed to a 0-100 scale. For functional scales and the global health status/QoL scale, higher scores represent better functioning or quality of life. For symptom scales/items, higher scores indicate more severe symptoms.
Lymphedema Surveillance (L-Dex Score) - (Lower SES) | Baseline to 3 Month Follow Up
  Change in L-Dex Score. Lymphedema surveillance will be completed using the SOZOs Bioimpedance device and monitored with the L-Dex score provided by the device. The L-Dex score is derived from bioimpedance spectroscopy measurements, which assess the resistance and reactance of body tissues to an electrical current. This provides detailed information about fluid levels in the body. The L-Dex score typically ranges from -10 to +10, with values outside this range indicating potential fluid accumulation and risk of lymphedema.
Lymphedema Surveillance (L-Dex Score) - (Higher SES) | Baseline to 3 Month Follow Up
  Change in L-Dex Score. Lymphedema surveillance will be completed using the SOZOs Bioimpedance device and monitored with the L-Dex score provided by the device. The L-Dex score is derived from bioimpedance spectroscopy measurements, which assess the resistance and reactance of body tissues to an electrical current. This provides detailed information about fluid levels in the body. The L-Dex score typically ranges from -10 to +10, with values outside this range indicating potential fluid accumulation and risk of lymphedema.
Lymphedema Surveillance (L-Dex Score) - Overall Change in Score | Baseline to 3 Month Follow Up
  Change in score of the L-Dex Score. Lymphedema surveillance will be completed using the SOZOs Bioimpedance device and monitored with the L-Dex score provided by the device. The L-Dex score is derived from bioimpedance spectroscopy measurements, which assess the resistance and reactance of body tissues to an electrical current. This provides detailed information about fluid levels in the body. The L-Dex score typically ranges from -10 to +10, with values outside this range indicating potential fluid accumulation and risk of lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Clark, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States